CLINICAL TRIAL: NCT05774769
Title: Commissural Closure to Treat Severe Mitral Regurgitation: Standing the Test of Time.
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: COSMIR
Record Dates: First submitted 2023-01-30; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Degenerative Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Commissural edge to edge mitral valve repair — Edge to edge is the suture of mitral valve leaflets tissue in the regurgitant spot. If the regurgitant jet is near a mitral commissure, it is called a commissural edge to edge.

SUMMARY:
Mitral regurgitation (MR) for degenerative disease is nowadays routinely treated with valve repair with excellent short and long term results in experienced centers. However, repair durability can varies according to the characteristics of the initial lesion, and better long term durability in isolated lesions of the posterior leaflets compared to anterior or bi-leaflets prolapse has been shown. A commissural MR can be caused by lesions of the anterior, posterior or both leaflets and several surgical techniques have been proposed to treat these lesions. However, long term outcomes of mitral valve repair (MVr) for isolated commissural flail or prolapse remain poor defined. In San Raffaele Hospital cardiac surgery, commissural lesions are usually treated with a functional approach, by means of edge-to-edge approximation of the anterior and posterior leaflet at the commissural area (commissural closure). The investigators previously reported the short and mid-term outcomes of this technique with satisfactory results. With this study the investigators aim to analyze the very long term clinical and echocardiographic results of isolated commissural lesions treated with commissural closure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Patients underwent mitral valve repair for flail or isolated commissural prolapse, of posterior, anterior or bileaflet origin;
* Patients operated on with median sternotomy or left minithoracotomy;
* Patients in whom the commissural MR has been treated with commissural closure and annuloplasty;
* Patients operated on at the Cardiac Surgery department of San Raffaele Hospital from January 1997 to December 2007.

Exclusion Criteria:

* Patients underwent a mitral valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a degenerative mitral valve disease in whom regurgitation occurred in commissural position, hence were treated with a commisural edge to edge surgery
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 14,5 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No